CLINICAL TRIAL: NCT02672033
Title: Neoadjuvant Accelerated Hypofractionated Radiation Therapy Immediately Prior to Radical Pleurectomy/Decortication for Malignant Pleural Mesothelioma: A Pilot Study
Brief Title: Accelerated Hypofractionated Radiation Therapy Immediately Before Surgery in Treating Patients With Malignant Pleural Mesothelioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-000487; NCI-2015-01736 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID552 (Other: Jonsson Comprehensive Cancer Center); 15-000487 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-11-02; First posted 2016-02-03 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-05

CONDITIONS: Pleural Epithelioid Mesothelioma; Pleural Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Radiation Dose Hypofractionation; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (hypofractionated IMRT, pleurectomy/decortication) (Experimental): Patients undergo 5 fractions of accelerated hypofractionated IMRT over 1 week with simultaneous integrated boost to gross disease. Patients then undergo pleurectomy/decortication within 14 days after completion of IMRT.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo accelerated hypofractionated IMRT
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Radiation: Intensity-Modulated Radiation Therapy — Undergo accelerated hypofractionated IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo pleurectomy/decortication

SUMMARY:
This pilot phase 0 trial studies accelerated hypofractionated radiation therapy immediately before surgery in treating patients with malignant pleural mesothelioma (cancer in the thin layer of tissue that covers the lungs and lines the interior wall of the chest cavity). Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Hypofractionated radiation therapy is a type of radiation therapy in which the total prescribed dose of radiation is divided into fewer but larger doses as compared to conventional radiation therapy. Giving accelerated hypofractionated radiation therapy immediately before surgery may improve survival, and may also reduce side effects experienced by patients with pleural mesothelioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and toxicity (both acute and chronic) of accelerated hypofractionated neoadjuvant helical intensity modulated radiation therapy prior to pleurectomy/decortication for malignant pleural mesothelioma.

SECONDARY OBJECTIVES:

I. To determine the pathologic complete response rate (pCR). II. To determine the tumor local control rate (LC). III. To determine the malignant pleural mesothelioma disease specific survival (DSS).

IV. To determine the overall survival (OS). V. To assess transforming growth factor beta (TGF-B), interleukin (IL)-1, and IL-6 levels as predictive biomarkers for treatment induced tissue injury.

VI. To assess the changes in the postoperative pleural immunological milieu in terms of chemo- and cytokine expression.

OUTLINE:

Patients undergo 5 fractions of accelerated hypofractionated intensity-modulated radiation therapy (IMRT) over 1 week with simultaneous integrated boost to gross disease. Patients then undergo pleurectomy/decortication within 14 days after completion of IMRT.

After completion of study treatment, patients are followed up at 6 weeks, and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelioid predominantly (> 70%) subtype malignant pleural mesothelioma
* Patient must have been evaluated by a University of California Los Angeles (UCLA) thoracic surgeon, and deemed medically and technically suitable for a pleurectomy/decortication procedure
* Karnofsky performance status (KPS) >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-2
* If a woman is of childbearing potential, a negative urine or serum pregnancy test must be documented; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study participation and for up to 4 weeks following the study

Exclusion Criteria:

* Patients who have previously received therapeutic radiation therapy to the chest
* Active systemic, pulmonary, or pericardial infection
* Use of chemotherapy within 4 weeks of the planned start of radiation therapy
* Pregnant women, or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period and for up to 4 weeks after the study
* Refusal to sign the informed consent
* Patients who are participating in a concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Percy Lee, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 10/2015 to 04/2018, 2 subjects were consented into the trial.
Pre-assignment Details: Eligibility screening by the Jonsson Comprehensive Cancer Center Data Safety Monitoring Board. Subjects undergo 5 fractions of hypofractionationated Intensity Modulated Radiation Therapy (IMRT) over 1 week with simultaneous integrated boost to gross disease.Subjects then undergo pleurectomy/decortication within 14 days after completion of IMRT.
Period: Overall Study
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  Age: 63 Years | 1
  Age: 69 Years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Ability to Accrue Sufficient Patients to Draw Conclusions About Endpoints in a Timely and Expedient Manner
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 1 year
Population: Data was not collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence of Acute and Subacute Toxicity Defined as Grade 4 or 5 Adverse Events as Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 3 months
Population: Data was not collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

3. Primary Outcome: Incidence of Chronic Toxicity as Assessed by the NCI CTCAE Version 4.0
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 5 years post-treatment
Population: Data was not collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

4. Secondary Outcome: Disease Specific Survival (DSS)
Description: Cumulative incidence approach will be used to estimate DSS. No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 5 years post-treatment
Population: No data was collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

5. Secondary Outcome: Local Control (LC)
Description: Cumulative incidence approach will be used to estimate the local failure rates. No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 5 years post-treatment
Population: No data was collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS)
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 5 years post-treatment
Population: Data was not collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

7. Secondary Outcome: Pathologic Complete Response Rate (pCR)
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 5 years post-treatment
Population: Data was not collected
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from 10/2015 until 4/2018, 30 months.
Description: Dose limiting toxicity (DLT) defined as any treatment-related grade 3 or higher toxicity in the following categories: respiratory, upper GI, and cardiac. Also, any other grade 4 or 5 toxicity attributed to the therapy constitutes DLT. All AE's and SAE's, with grade and attribution were submitted to our DSMB as part of our quarterly summary reports. Serious adverse events were also reported individually to the DSMB and, where required, to our UCLA IRB within 2-10 days of awareness.
Arm/Group | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication)
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication) (N=2)
Death (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Expired from respiratory failure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated IMRT, Pleurectomy/Decortication) (N=2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weakness (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the rarity of malignant pleural mesothelioma only two patients were enrolled and treated. There number as insufficient for any analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes